CLINICAL TRIAL: NCT01776190
Title: Low-dose UVA1 Radiation in Cutaneous Lupus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben Chong (Other)
Collaborators: Daavlin Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ben Chong, Associate Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072012-024
Record Dates: First submitted 2012-08-30; First posted 2013-01-28 (Estimated); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UVA1 treatment (Experimental): Low-dose UVA1 will be applied to active cutaneous lupus lesions three times a week for 10 weeks.
  Interventions: Device: UVA1 radiation treatment

INTERVENTIONS:
Device: UVA1 radiation treatment

SUMMARY:
The investigators are conducting an open-label clinical trial determining the effects of UVA1 phototherapy on cutaneous lupus (CLE) patients. Past research on systemic lupus (SLE) subjects indicates that this treatment is likely to be effective in treating cutaneous lupus with few side effects. The fact that most CLE patients are seen at dermatology clinics also increases the usefulness of this study because there is a large probability that phototherapy treatment will be accessible for many of the patients that stand to benefit from it.

DETAILED DESCRIPTION:
Study subjects will receive low dose (20 J/cm2) UVA1 phototherapy treatment three times per week for 10 weeks. Each treatment will take less than 30 minutes. This period will be followed by an eight-week observation phase to assess longer term effects of the treatment. Patients will be assessed for disease activity, and blood studies and photos will be completed prior to, during, and after phototherapy treatment. Optional skin biopsies of affected and unaffected skin will be performed at the beginning and end of the active treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* You must be 18 years or older with a diagnosis of cutaneous lupus.
* You must have at least two active areas of cutaneous lupus.
* You will need to come in three days a week for a 10-week period.
* You will need to participate in four physician visits and blood draws.

Exclusion Criteria:

* You do not have a diagnosis of cutaneous lupus.
* You have less than two active areas of cutaneous lupus.
* You are unable to come in three days a week for treatment for a 10-week period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin F Chong, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- UVA1 Treatment: Low-dose UVA1 will be applied to active cutaneous lupus lesions three times a week for 10 weeks.
  UVA1 radiation treatment
Period: Overall Study
Arm/Group | UVA1 Treatment
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | UVA1 Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [30.8 to 49.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) Activity Score
Description: The CLASI activity score represents the amount of skin disease activity in cutaneous lupus patients, as evaluated by a provider. The minimum score is 0 (no disease activity), and the maximum score is 70 (maximum/worst disease activity). The change is measured at the start and end of the UVA1 trial therapy.
Time Frame: 10 weeks
Population: Cutaneous Lupus Erythematosus patients
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | UVA1 Treatment
Number analyzed (Participants) | 5
Units on a scale | -1 [-1 to 1]

2. Secondary Outcome: Change in Cutaneous Lupus Disease Area and Severity Index (CLASI) Damage Score
Description: The CLASI damge score represents the amount of skin disease damage in cutaneous lupus patients, as evaluated by a provider. The minimum score is 0 (no disease damage), and the maximum score is 80 (maximum/worst disease damage). The change is measured at the start and end of the UVA1 trial therapy.
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | UVA1 Treatment
Number analyzed (Participants) | 5
Units on a scale | 0 [0 to 2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 18 week observation period for each patient.
Arm/Group | UVA1 Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Limitations include small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT01776190/Prot_SAP_000.pdf